CLINICAL TRIAL: NCT04674046
Title: Deep Deltoid Ligament Integrity in Ankles With Isolated Weber Type B Fractures - Mini-invasive Arthroscopic Evaluation Using the Arthrex NanoScope.
Brief Title: Deep Deltoid Ligament Integrity in Weber B Ankle Fractures - Mini-invasive Arthroscopic Evaluation.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ostfold Hospital Trust (Other)
Responsible Party: Principal Investigator, Marius Molund, Senior Consultant Foot and Ankle Surgery, Ostfold Hospital Trust
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 123245
Record Dates: First submitted 2020-11-17; First posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Ankle Fracture - Lateral Malleolus; Deltoid Ligament; Sprain (Strain) (Ankle); Ankle Fractures
Keywords: Weber B; Rotational ankle fracture; Ankle stability; Deep deltoid ligament; Deltoid ligament injury
MeSH Terms: conditions — Ankle Fractures; Sprains and Strains | interventions — Conservative Treatment; Open Fracture Reduction; Fracture Fixation, Internal

STUDY DESIGN:
Intervention Model Description: Prospective cohort study where participants will be assigned to nonoperative or operative treatment based on minimally invasive arthroscopic evaluation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nonoperative treatment if deltoid ligament is intact (Experimental): AirCast Air-stirrup (DJO Global) functional orthosis for 6 weeks.
  Interventions: Device: Nonoperative treatment; Behavioral: Standardized education
- Operative treatment if deltoid ligament is ruptured (Experimental): Open reduction, internal fixation of the fibular fracture using plate and screws.
  Interventions: Procedure: Operative treatment; Behavioral: Standardized education

INTERVENTIONS:
Device: Nonoperative treatment — Patients where the ankle is evaluated as stable using arthroscopy will be treated with conservative treatment using a functional brace (AirCast) for 6 weeks. Participants will be instructed to bear weight as tolerated and to actively do standardized range-of-motion exercises.
  Other Names: Conservative Treatment
  Arms: Nonoperative treatment if deltoid ligament is intact
Procedure: Operative treatment — Patients where the ankle is evaluated as unstable using arthroscopy will be operated on. Standard operative treatment is open reduction and internal fixation (ORIF) of the fracture using plate and screws. The goal is an osteosynthesis that allow for early range-of-motion exercises, but weightbearing is usually not tolerated until 6 weeks postoperatively.
  Other Names: Open reduction, internal fixation
  Arms: Operative treatment if deltoid ligament is ruptured
Behavioral: Standardized education — All participants, regardless of group allocation, will receive education focusing on basic self- management. A physiotherapist will be responsible for the education. The intention will be to increase self-efficacy and encourage self-management. Participants will learn about crutch walking, cast or orthosis usage, loading principles, be advised to stay physically active within proper restrictions and how to rest and reduce pain and swelling of the ankle in the acute phase. Participants will also receive a standard information brochure about the condition, treatment and basic self-management.

SUMMARY:
Prospective cohort study to evaluate the use of a NanoScopic procedure to assess deltoid ligament injuries with outcomes measured at baseline, 6 weeks, 12 weeks, 1 year and 2 years. Further to examine whether the findings correlate with results on gravity stress test and weightbearing radiographs.

DETAILED DESCRIPTION:
Purpose and research question The main purpose is to evaluate integrity in the deep deltoid ligament in ankles with isolated Weber type B fractures using a minimally invasive Nanoscopic technique. Further results of a Nanoscopic evaluation will be correlated to the results of gravity stress and weightbearing radiographs. Additionally, the Nanoscopic evaluation will be used to assess associated injuries including cartilage and syndesmotic lesions.

Methods Primary evaluation will be done in the acute setting. All isolated Weber type B fractures without radiological signs of instability (medial clear space of 7 mm or less) on initial non-weightbearing radiographs presenting to our clinic will be evaluated for inclusion. Nanoscopic evaluation will determine stability for all patients with radiographic measurements indicating "uncertain stability". "Uncertain stability" of the ankle is assumed when at least one out of 3 (plain-, gravity- or weightbearing-) radiographs is showing instability. Like Seidel et al. (2017), in the event of a MCS of over 7 mm on initial non-weightbearing radiographs the ankle is considered unstable and will be evaluated for surgery. These patients will not be evaluated for inclusion.

For radiographic tests the size of the MCS will make up an indirect measurement of deltoid ligament capacity. The MCS is defined as the distance between the medial border of the talus and the lateral border of the medial malleolus on a line parallel to and 5 mm below the talar dome on anteroposterior radiographs. A MCS of 5 mm or less defines the ankle as stable. An MCS >5 mm AND 1 mm or more increase compared to the contralateral (non-injured ankle) ankle defines the ankle as unstable.

Plain-, weightbearing- and gravity stress radiographs and nanoscopic evaluation will be done 3-14 days after injury at the outpatient clinic. The radiographic test battery will be done prior to nanoscopy. Only patients demonstrating at least one positive stress radiograph (weightbearing or gravity) or a plain radiograph with a MCS measurement above the threshold (5 mm AND 1 mm or more increase compared to the contralateral ankle) will undergo nanoscopic evaluation.

Participants with "uncertain" stability will be assigned to non-operative or surgical treatment based on ankle stability evaluation using results from the NanoScopic evaluation consistently. Stability is assumed when the posterior part of the deep deltoid ligament is visible and intact. Stable ankles will be treated non-operatively with a functional brace (AirCast) for 6 weeks. Participants will be instructed to bear weight as tolerated and to actively do standardized range-of-motion exercises. Unstable ankles will be operated on. Standard operative treatment is open reduction and internal fixation of the fracture using plate and screws. The goal is an osteosynthesis that allow for early range-of-motion exercises, but weightbearing is usually not tolerated until 6 weeks postoperatively.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* With isolated Weber type B fractures without radiological signs of medial clear space widening on initial plain radiographs (MCS < 7mm).
* Demonstrating at least one positive stress radiograph (weightbearing or gravity) or a plain radiograph with a MCS measurement above the threshold (5 mm AND 1 mm or more increase compared to the contralateral ankle) (WP2).
* 18-80 years of age.
* With pre-injury walking ability without aids.

Exclusion Criteria:

Patients:

* With fracture of the medial malleolus, pre-hospital closed fracture reduction, open fracture, fracture resulting from high-energy trauma or multi-trauma and pathologic fracture.
* With poorly regulated Diabetes Mellitus type 1 and 2, neuropathies and generalized joint disease such as Rheumatoid Arthritis.
* That are assumed not compliant (drug use, cognitive- and/or psychiatric disorders).
* With previous history of ipsilateral ankle fracture.
* With previous history of ipsilateral major ankle-/foot surgery.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-09-15 (Actual); Primary Completion 2024-09-15 (Estimated); Study Completion 2024-09-15 (Estimated)

PRIMARY OUTCOMES:
Change in Manchester-Oxford Foot Questionnaire (MOXFQ) | 6 weeks, 12 weeks, 52 weeks, 104 weeks
  The MOXFQ (Dawson et al., 2006) was developed to measure perceived foot- specific functioning and health-related quality of life. The MOXFQ is supported as the current most valid, reliable and responsive ankle-specific instrument (Jia, Huang, & Gagnier, 2017) and has been validated for use in ankle pathology (Dawson et al., 2011). It is available in Norwegian, but it has not been validated in its translated form. The score comprises a total of 16 items. They are distributed within 3 dimensions; foot pain (5 items), walking/standing (7 items) and social interaction (4 items) where all items are scored on a 5-point Likert scale, scored 0 (best) to 4 (worst). The MOXFQ index (Morley et al., 2013) will be used, where scores are converted to a metric (0-100) scale. Lower scores indicate less pain and higher levels of ankle/foot functioning (Morley et al., 2013).

SECONDARY OUTCOMES:
Registration of adverse events | 104 weeks.
  Adverse events including malalignment, deep vein trobosis, nerve injury, wound infection, delayed wound healing and crossover to surgery (including reason for crossover).
Registration of fracture union | 12 weeks.
  Fracture union will be registered as union/nonunion and defined as concurrent radiographic evidence of fracture union and pain-free palpation over the fracture location.
Registration of the incidence of concomitant cartilage injuries. | Baseline.
  Evaluated peroperatively by minimally invasive arthroscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Marius Molund, Md, PhD, Principal Investigator — Ostfold HT
Locations (1):
- Østfold HT, Sarpsborg, Østfold fylke, Norway

IPD SHARING:
Plan to Share IPD: No